CLINICAL TRIAL: NCT01009554
Title: Assessment of the Oral Tissue Tolerance of a Potassium Oxalate Containing Mouthrinse
Brief Title: Oral Tissue Tolerance of a Mouthrinse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UNKPLT0002
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Dental Health
Keywords: Mouthwashes
MeSH Terms: interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Potassium Oxylate (Experimental): 1.5% potassium oxalate sensitive mouthwash
  Interventions: Device: Potassium Oxylate Mouthwash
- Sodium Fluoride (Active Comparator): Sodium Fluoride Dentifrice
  Interventions: Drug: Sodium Fluoride Dentifrice

INTERVENTIONS:
Device: Potassium Oxylate Mouthwash — Rinse with 10 mL for 60 seconds, twice daily after brushing in usual manner with a sodium fluoride dentifrice
  Other Names: Formula 11794-050
  Arms: Potassium Oxylate
Drug: Sodium Fluoride Dentifrice — Brush in usual manner, twice daily, with a sodium fluoride dentifrice
  Other Names: Regular Cavity Protection toothpaste
  Arms: Sodium Fluoride

SUMMARY:
This study is 8 weeks long. People participating in this study will be asked to brush their teeth two times a day. Some people will get a mouthwash. People with a mouthwash will rinse two times a day after brushing their teeth. The mouth, teeth, tongue and gums will be looked at by a dentist. The dentist will look at the mouth to make sure the mouthwash does not irritate the mouth. The dentist will also look at the color of the teeth and amount of stain on the front teeth.

DETAILED DESCRIPTION:
This is an 8-week, randomized, observer-blind, controlled, parallel group clinical study design to assess the oral tissue tolerance of a potassium oxalate containing mouthrinse. Subjects will have their oral soft/hard tissues assessed and will be evaluated for stain levels and tooth color shades at Screening/Baseline (Visit 1), Week 4 (Visit 2), Week 6 (Visit 3) and Week 8 (Visit 4). Subjects will be instructed to brush their teeth two times daily in their usual manner using the provided sodium fluoride toothpaste. Subjects assigned to the mouthrinse group will be instructed to rinse twice daily after brushing.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age and in good general and oral health.
* Volunteers must read, sign, and receive a signed copy of the Informed Consent Form after the nature of the study has been fully explained.
* Willingness to use the assigned products according to instructions, availability for appointments and likelihood of completing the study.
* Willingness to refrain from using any breath freshener products or unassigned oral care products (i.e., oral care strips, candy-type mints, sprays, chewing gums, throat lozenges, cough drops, mouthwashes or teeth whitening products) throughout the duration of the study.
* Willingness to refrain from using any whitening products and smokeless tobacco products within one week prior to and for the duration of the study, in order to reduce alternate sources of potential irritation.
* A minimum of 16 natural teeth, including at least 10 of the 12 anterior teeth (#6-11, #22-27, however, #7-10 must be present), with scorable facial and lingual surfaces. Teeth that are grossly carious, fully crowned or extensively restored on facial and/or lingual surfaces, orthodontically banded, abutments, or third molars will not be included in the tooth count.
* Classic Vita® Shade minimum value of A2 or darker on at least 2 of the 4 maxillary anterior teeth (#7-10).
* Absence of abnormal or severely fissured tongue, geographic tongue, tongue piercing or any obvious tongue abnormalities that may interfere with the assessment of oral irritation.
* Adequate oral hygiene (i.e., brush teeth daily and exhibit no signs of oral neglect).
* Absence of neglected dental health (i.e. gross calculus deposits or rampant caries based on visual examination), significant oral soft tissue pathology, systemically-related gingival enlargement, tissue damage due to ill-fitting appliances or restoration, or extreme crowding or overlapping of teeth

Exclusion Criteria:

* Physical limitations or restrictions that might preclude use of normal oral hygiene procedures (i.e., toothbrushing, etc.).
* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses.
* History or current evidence of significant oral soft tissue pathology, excluding gingivitis, based on the dentist's visual examination and at the discretion of the investigator.
* Prior participation in any oral hygiene or product clinical study within the previous 30 days.
* Therapy with any medications, currently or within the last 30 days, which might interfere with the outcome of the study by affecting tooth color or stain formation (i.e., certain antimicrobial mouthrinses and antibiotics, such as chlorhexidine).
* Restorations on 10% or more of the facial surfaces of the maxillary anterior incisor teeth.
* Dental fluorosis, hypoplasia, restorations, tetracycline stains, or other enamel surface irregularities that may interfere with evaluation of the selected teeth.
* Visual evidence of Moderate/advanced periodontitis (ADA Type III, IV). Orthodontic bands, appliances, bridges, numerous crowns, removable orthodontic appliances or partial dentures.
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results).
* Regular use of whitening products within 1 week prior to Screening/Baseline. Other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial result and, in the judgment of the investigator, would make the subject inappropriate for the entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lynch, DMD, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- TKL Reearch, Inc., Paramus, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Crest® Regular Toothpaste: Crest® Cavity Protection Regular Toothpaste (Brushing Only)
- 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse): Crest® Cavity Protection followed by 1.5% Potassium Oxalate & pH 4.2 Mouth Rinse (Brushing followed by Mouth Rinse)
Period: Overall Study
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Started | 48 | 48
Completed | 46 | 41
Not Completed | 2 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Noncompliant with Study Product | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse) | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.96) | 49.8 (8.08) | 48.7 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  USA | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Tooth Color as Represented by ΔE at 8 Weeks Post Baseline From the CIElab Assessment
Description: The tooth color of the four maxillary incisor teeth (teeth #7-10, facial surface) was measured instrumentally using the MHT SpectroShade System. Assessments were made under standardized lighting conditions after participants brushed their teeth with water. The aperture tip was placed perpendicularly to the facial surface of the tooth and the color measured using the CIElab color system. The changes in the individual L*, a*, and b* color parameters were calculated to determine quantitatively the improvements in tooth lightness, redness, and yellowness, respectively. An overall change in tooth color was calculated using the CIE color equation ΔE = [(ΔL*)^2 + (Δa*)^2 + (Δb*)^2]^1/2. The ΔE was calculated per tooth and then averaged over the teeth for a participant.
Time Frame: 8 weeks
Population: Analysis was based on the Full Analysis Set, defined as all randomized participants who used the investigational product and had baseline and at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.909 (0.0612) | 1.035 (0.0650)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); The null hypothesis was no difference in mean outcome between treatment groups. The alternative hypothesis was a difference in mean outcome between treatment groups; Test type: Superiority or Other; p = 0.168, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline tooth color parameter values (L, a, and b) and age (in years) as covariates; Least Squares Mean Difference = 0.126, 95% CI 2-sided [-0.054 to 0.306], Standard Error of Mean 0.0905

2. Primary Outcome: Oral Tissue Tolerance
Description: Oral tissue tolerance was assessed by oral tissue adverse events for which the relationship to treatment was considered as possible, probable, or very likely. If the relationship to treatment was missing, the adverse event was categorized as a treatment-related adverse event.
Time Frame: through 8 weeks
Population: Analysis was based on the Safety Analysis Set, defined as all participants who used at least one dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 48 | 48
percentage of participants
  Participants with ≥ one treatment-related AE | 2.1 | 0.0
  Sensitivity of teeth | 2.1 | 0.0

3. Secondary Outcome: Change in Tooth Color as Represented by ΔE at 4 Weeks Post Baseline From the CIElab Assessment
Description: as for outcome 1
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.875 (0.0464) | 0.882 (0.0475)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.928, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.006, 95% CI 2-sided [-0.127 to 0.139], Standard Error of Mean 0.0670

4. Secondary Outcome: Change in Tooth Color as Represented by ΔE at 6 Weeks Post Baseline From the CIElab Assessment
Description: as for outcome 1
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.805 (0.0496) | 1.040 (0.0507)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.235, 95% CI 2-sided [0.092 to 0.378], Standard Error of Mean 0.0718

5. Secondary Outcome: Change in Tooth Color as Represented by ΔL at 4 Weeks Post Baseline From the CIElab Assessment
Description: The tooth color of the four maxillary incisor teeth (teeth #7-10, facial surface) was measured instrumentally using the MHT SpectroShade System. Assessments were made under standardized lighting conditions after participants brushed their teeth with water. The aperture tip was placed perpendicularly to the facial surface of the tooth and the color measured using the CIElab color system. The change in the individual L* color parameter was calculated. The ΔL was calculated per tooth and then averaged over the teeth for a participant.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.013 (0.0857) | 0.054 (0.0876)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.741, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline tooth color parameter value L and age (in years) as covariates; Least Squares Mean Difference = 0.041, 95% CI 2-sided [-0.205 to 0.286], Standard Error of Mean 0.1235

6. Secondary Outcome: Change in Tooth Color as Represented by ΔL at 6 Weeks Post Baseline From the CIElab Assessment
Description: as for outcome 5
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.071 (0.0959) | -0.090 (0.0981)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.249, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline tooth color parameter value L and age (in years) as covariates; Least Squares Mean Difference = -0.161, 95% CI 2-sided [-0.437 to 0.115], Standard Error of Mean 0.1386

7. Secondary Outcome: Change in Tooth Color as Represented by ΔL at 8 Weeks Post Baseline From the CIElab Assessment
Description: as for outcome 5
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.158 (0.0949) | -0.043 (0.1006)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.154, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline tooth color parameter value L and age (in years) as covariates; Least Squares Mean Difference = -0.201, 95% CI 2-sided [-0.479 to 0.077], Standard Error of Mean 0.1398

8. Secondary Outcome: Change in Tooth Color as Represented by Δb at 4 Weeks Post Baseline From the CIElab Assessment
Description: The tooth color of the four maxillary incisor teeth (teeth #7-10, facial surface) was measured instrumentally using the MHT SpectroShade System. Assessments were made under standardized lighting conditions after participants brushed their teeth with water. The aperture tip was placed perpendicularly to the facial surface of the tooth and the color measured using the CIElab color system. The change in the individual b* color parameter was calculated. The Δb was calculated per tooth and then averaged over the teeth for a participant.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.077 (0.0518) | -0.117 (0.0529)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.011, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline tooth color parameter value b and age (in years) as covariates; Least Squares Mean Difference = -0.195, 95% CI 2-sided [-0.343 to -0.047], Standard Error of Mean 0.0746

9. Secondary Outcome: Change in Tooth Color as Represented by Δb at 6 Weeks Post Baseline From the CIElab Assessment
Description: as for outcome 8
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.123 (0.0487) | -0.212 (0.0498)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline tooth color parameter value b and age (in years) as covariates; Least Squares Mean Difference = -0.334, 95% CI 2-sided [-0.474 to -0.195], Standard Error of Mean 0.0703

10. Secondary Outcome: Change in Tooth Color as Represented by Δb at 8 Weeks Post Baseline From the CIElab Assessment
Description: as for outcome 8
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.107 (0.0639) | -0.107 (0.0677)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.025, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline tooth color parameter value b and age (in years) as covariates; Least Squares Mean Difference = -0.214, 95% CI 2-sided [-0.401 to -0.027], Standard Error of Mean 0.0939

11. Secondary Outcome: Mean Stain Score Over All Tooth Sites at 4 Weeks
Description: The mean stain score (0-9) per participant was determined by multiplying the individual area and intensity scores from each region and summing them then dividing by the number of sites scored. The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). All four regions were scored for area and intensity according to the following criteria. Stain area for mesial, gingival, and distal regions were scored on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain covers entire area) and for the body of tooth on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain outside pits/grooves, over 10% of surface affected). The intensity of yellow-brown stains occurring in each region was assessed on a 4-point ordinal scale (0=no stain; 3=heavy, dark stain).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.329 (0.0464) | 0.386 (0.0505)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.319, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain score over all tooth sites and smoking status as covariates; Least Squares Mean Difference = 0.056, 95% CI 2-sided [-0.055 to 0.168], Standard Error of Mean 0.0562

12. Secondary Outcome: Mean Stain Score Over All Tooth Sites at 6 Weeks
Description: as for outcome 11
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.349 (0.0565) | 0.621 (0.0605)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 11, analysis 1]; Least Squares Mean Difference = 0.272, 95% CI 2-sided [0.139 to 0.405], Standard Error of Mean 0.0668

13. Secondary Outcome: Mean Stain Score Over All Tooth Sites at 8 Weeks
Description: as for outcome 11
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.394 (0.0703) | 0.791 (0.0785)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 11, analysis 1]; Least Squares Mean Difference = 0.398, 95% CI 2-sided [0.231 to 0.565], Standard Error of Mean 0.0840

14. Secondary Outcome: Mean Stain Intensity Over All Tooth Sites at 4 Weeks
Description: The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). All four regions were scored for intensity according to the following criteria. The intensity of yellow-brown stains occurring in each region is unrelated to the area covered with stained pellicle. All four regions were assessed on a 4-point ordinal scale as 0=no stain, 1=faint stain (can be seen with close examination), 2=moderate stain (clearly visible and aesthetically unacceptable), 3=heavy, dark stain (obvious and aesthetically unacceptable).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.154 (0.0224) | 0.184 (0.0243)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.270, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain intensity over all tooth sites and smoking status as covariates; Least Squares Mean Difference = 0.030, 95% CI 2-sided [-0.024 to 0.084], Standard Error of Mean 0.0271

15. Secondary Outcome: Mean Stain Intensity Over All Tooth Sites at 6 Weeks
Description: as for outcome 14
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.164 (0.0274) | 0.302 (0.0293)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 14, analysis 1]; Least Squares Mean Difference = 0.137, 95% CI 2-sided [0.073 to 0.202], Standard Error of Mean 0.0324

16. Secondary Outcome: Mean Stain Intensity Over All Tooth Sites at 8 Weeks
Description: as for outcome 14
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.181 (0.0334) | 0.375 (0.0372)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 14, analysis 1]; Least Squares Mean Difference = 0.193, 95% CI 2-sided [0.114 to 0.273], Standard Error of Mean 0.0399

17. Secondary Outcome: Mean Stain Area Over All Tooth Sites at 4 Weeks
Description: The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). All four regions were scored for area according to the following criteria. Stain area for mesial, gingival, and distal regions were scored as 0=no stain present, natural tooth color; 1=thin line of stain, may be discontinuous; 2=thick line or band of stain; 3=stain covers entire area and for the body of tooth as 0=no stain present, natural tooth color, 1=stain limited to pits and grooves; 2=stain outside pits/grooves, up to 10% of surface affected; 3=stain outside pits/grooves, over 10% of surface affected.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.162 (0.0225) | 0.196 (0.0245)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.217, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area over all tooth sites and smoking status as covariates; Least Squares Mean Difference = 0.034, 95% CI 2-sided [-0.020 to 0.088], Standard Error of Mean 0.0273

18. Secondary Outcome: Mean Stain Area Over All Tooth Sites at 6 Weeks
Description: as for outcome 17
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.166 (0.0270) | 0.303 (0.0290)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area over all tooth sites and smoking status as covariates; Least Squares Mean Difference = 0.137, 95% CI 2-sided [0.073 to 0.200], Standard Error of Mean 0.0320

19. Secondary Outcome: Mean Stain Area Over All Tooth Sites at 8 Weeks
Description: as for outcome 17
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.188 (0.0340) | 0.383 (0.0379)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area over all tooth sites and smoking status as covariates; Least Squares Mean Difference = 0.195, 95% CI 2-sided [0.114 to 0.276], Standard Error of Mean 0.0406

20. Secondary Outcome: Mean Stain Score for Interproximal (Mesial and Distal) Sites at 4 Weeks
Description: The mean stain score (0-9) per participant was determined by multiplying the individual area and intensity scores from each region and summing them then dividing by the number of sites scored. The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). Stain area for mesial and distal regions were scored on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain covers entire area). The intensity of yellow-brown stains occurring in each region was assessed on a 4-point ordinal scale (0=no stain; 3=heavy, dark stain).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.408 (0.0590) | 0.463 (0.0643)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.444, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area score for interproximal (mesial and distal) sites and smoking status as covariates; Least Squares Mean Difference = 0.055, 95% CI 2-sided [-0.087 to 0.197], Standard Error of Mean 0.0716

21. Secondary Outcome: Mean Stain Score for Interproximal (Mesial and Distal) Sites at 6 Weeks
Description: as for outcome 20
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.427 (0.0712) | 0.776 (0.0762)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain score for interproximal (mesial and distal) sites and smoking status as covariates; Least Squares Mean Difference = 0.349, 95% CI 2-sided [0.182 to 0.517], Standard Error of Mean 0.0843

22. Secondary Outcome: Mean Stain Score for Interproximal (Mesial and Distal) Sites at 8 Weeks
Description: as for outcome 20
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.451 (0.0889) | 0.994 (0.0991)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 21, analysis 1]; Least Squares Mean Difference = 0.542, 95% CI 2-sided [0.331 to 0.754], Standard Error of Mean 0.1063

23. Secondary Outcome: Mean Stain Intensity For Interproximal (Mesial and Distal) Sites at 4 Weeks
Description: The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). The interproximal (mesial and distal) regions were scored for intensity according to the following criteria. The intensity of yellow-brown stains occurring in each region is unrelated to the area covered with stained pellicle. The regions were assessed on a 4-point ordinal scale as 0=no stain, 1=faint stain (can be seen with close examination), 2=moderate stain (clearly visible and aesthetically unacceptable), 3=heavy, dark stain (obvious and aesthetically unacceptable).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.192 (0.0284) | 0.224 (0.0309)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.361, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain intensity for interproximal (mesial and distal) sites and smoking status as covariates; Least Squares Mean Difference = 0.032, 95% CI 2-sided [-0.037 to 0.100], Standard Error of Mean 0.0344

24. Secondary Outcome: Mean Stain Intensity For Interproximal (Mesial and Distal) Sites at 6 Weeks
Description: as for outcome 23
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.205 (0.0350) | 0.379 (0.0374)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = 0.174, 95% CI 2-sided [0.092 to 0.256], Standard Error of Mean 0.0414

25. Secondary Outcome: Mean Stain Intensity For Interproximal (Mesial and Distal) Sites at 8 Weeks
Description: as for outcome 23
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.210 (0.0422) | 0.475 (0.0470)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 23, analysis 1]; Least Squares Mean Difference = 0.264, 95% CI 2-sided [0.164 to 0.364], Standard Error of Mean 0.0504

26. Secondary Outcome: Mean Stain Area for Interproximal (Mesial and Distal) Sites at 4 Weeks
Description: The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). The interproximal (mesial and distal) regions were scored for area according to the following criteria. Stain area for mesial and distal regions were scored as 0=no stain present, natural tooth color; 1=thin line of stain, may be discontinuous; 2=thick line or band of stain; 3=stain covers entire area.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.202 (0.0284) | 0.236 (0.0309)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.331, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area for interproximal (mesial and distal) sites and smoking status as covariates; Least Squares Mean Difference = 0.034, 95% CI 2-sided [-0.035 to 0.102], Standard Error of Mean 0.0345

27. Secondary Outcome: Mean Stain Area for Interproximal (Mesial and Distal) Sites at 6 Weeks
Description: as for outcome 26
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.206 (0.0348) | 0.383 (0.0373)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 26, analysis 1]; Least Squares Mean Difference = 0.177, 95% CI 2-sided [0.095 to 0.259], Standard Error of Mean 0.0414

28. Secondary Outcome: Mean Stain Area for Interproximal (Mesial and Distal) Sites at 8 Weeks
Description: as for outcome 26
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.218 (0.0433) | 0.483 (0.0483)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 26, analysis 1]; Least Squares Mean Difference = 0.265, 95% CI 2-sided [0.162 to 0.368], Standard Error of Mean 0.0519

29. Secondary Outcome: Mean Stain Score for Gingival Sites at 4 Weeks
Description: The mean stain score (0-9) per participant was determined by multiplying the individual area and intensity scores from each region and summing them then dividing by the number of sites scored. The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). Stain area for gingival regions were scored on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain covers entire area) and for the body of tooth on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain outside pits/grooves, over 10% of surface affected). The intensity of yellow-brown stains occurring in each region was assessed on a 4-point ordinal scale (0=no stain; 3=heavy, dark stain).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.383 (0.0596) | 0.521 (0.0652)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.060, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain score for the gingival region and smoking status as covariates; Least Squares Mean Difference = 0.138, 95% CI 2-sided [-0.006 to 0.282], Standard Error of Mean 0.0726

30. Secondary Outcome: Mean Stain Score for Gingival Sites at 6 Weeks
Description: as for outcome 29
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.395 (0.0732) | 0.732 (0.0786)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 29, analysis 1]; Least Squares Mean Difference = 0.338, 95% CI 2-sided [0.165 to 0.510], Standard Error of Mean 0.0870

31. Secondary Outcome: Mean Stain Score for Gingival Sites at 8 Weeks
Description: as for outcome 29
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.526 (0.0914) | 0.920 (0.1023)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 29, analysis 1]; Least Squares Mean Difference = 0.394, 95% CI 2-sided [0.176 to 0.612], Standard Error of Mean 0.1095

32. Secondary Outcome: Mean Stain Intensity for Gingival Sites at 4 Weeks
Description: The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). The gingival regions were scored for intensity according to the following criteria. The intensity of yellow-brown stains occurring in each region is unrelated to the area covered with stained pellicle. The gingival regions were assessed on a 4-point ordinal scale as 0=no stain, 1=faint stain (can be seen with close examination), 2=moderate stain (clearly visible and aesthetically unacceptable), 3=heavy, dark stain (obvious and aesthetically unacceptable).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.180 (0.0292) | 0.252 (0.0318)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.045, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain intensity for the gingival region and smoking status as covariates; Least Squares Mean Difference = 0.072, 95% CI 2-sided [0.002 to 0.143], Standard Error of Mean 0.0355

33. Secondary Outcome: Mean Stain Intensity for Gingival Sites at 6 Weeks
Description: as for outcome 32
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.180 (0.0350) | 0.358 (0.0375)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 32, analysis 1]; Least Squares Mean Difference = 0.178, 95% CI 2-sided [0.095 to 0.260], Standard Error of Mean 0.0415

34. Secondary Outcome: Mean Stain Intensity for Gingival Sites at 8 Weeks
Description: as for outcome 32
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.241 (0.0434) | 0.438 (0.0485)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 32, analysis 1]; Least Squares Mean Difference = 0.197, 95% CI 2-sided [0.094 to 0.300], Standard Error of Mean 0.0520

35. Secondary Outcome: Mean Stain Area for Gingival Sites at 4 Weeks
Description: The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). The gingival regions were scored for area according to the following criteria. Stain area for gingival regions were scored as 0=no stain present, natural tooth color; 1=thin line of stain, may be discontinuous; 2=thick line or band of stain; 3=stain covers entire area.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.186 (0.0292) | 0.263 (0.0319)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.034, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area for the gingival region and smoking status as covariates; Least Squares Mean Difference = 0.077, 95% CI 2-sided [0.006 to 0.147], Standard Error of Mean 0.0355

36. Secondary Outcome: Mean Stain Area for Gingival Sites at 6 Weeks
Description: as for outcome 35
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.184 (0.0335) | 0.352 (0.0359)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 35, analysis 1]; Least Squares Mean Difference = 0.168, 95% CI 2-sided [0.089 to 0.247], Standard Error of Mean 0.0398

37. Secondary Outcome: Mean Stain Area for Gingival Sites at 8 Weeks
Description: as for outcome 35
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.250 (0.0430) | 0.444 (0.0481)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 35, analysis 1]; Least Squares Mean Difference = 0.193, 95% CI 2-sided [0.091 to 0.296], Standard Error of Mean 0.0516

38. Secondary Outcome: Mean Stain Score for Body Sites at 4 Weeks
Description: The mean stain score (0-9) per participant was determined by multiplying the individual area and intensity scores from each region and summing them then dividing by the number of sites scored. The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). Stain area for the body of the tooth was scored on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain outside pits/grooves, over 10% of surface affected). The intensity of yellow-brown stains occurring in each region was assessed on a 4-point ordinal scale (0=no stain; 3=heavy, dark stain).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.132 (0.0258) | 0.112 (0.0281)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.524, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain score for the body region and smoking status as covariates; Least Squares Mean Difference = -0.020, 95% CI 2-sided [-0.082 to 0.042], Standard Error of Mean 0.0310

39. Secondary Outcome: Mean Stain Score for Body Sites at 6 Weeks
Description: as for outcome 38
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.160 (0.0337) | 0.215 (0.0361)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.172, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain score for the body region and smoking status as covariates; Least Squares Mean Difference = 0.055, 95% CI 2-sided [-0.024 to 0.133], Standard Error of Mean 0.0395

40. Secondary Outcome: Mean Stain Score for Body Sites at 8 Weeks
Description: as for outcome 38
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.143 (0.0371) | 0.258 (0.0412)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.010, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain score for the body region and smoking status as covariates; Least Squares Mean Difference = 0.116, 95% CI 2-sided [0.028 to 0.203], Standard Error of Mean 0.0439

41. Secondary Outcome: Mean Stain Intensity for Body Sites at 4 Weeks
Description: The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). The body regions were scored for intensity according to the following criteria. The intensity of yellow-brown stains occurring in each region is unrelated to the area covered with stained pellicle. The body regions were assessed on a 4-point ordinal scale as 0=no stain, 1=faint stain (can be seen with close examination), 2=moderate stain (clearly visible and aesthetically unacceptable), 3=heavy, dark stain (obvious and aesthetically unacceptable).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.058 (0.0121) | 0.045 (0.0132)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.348, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain intensity for the body region and smoking status as covariates; Least Squares Mean Difference = -0.014, 95% CI 2-sided [-0.043 to 0.015], Standard Error of Mean 0.0145

42. Secondary Outcome: Mean Stain Intensity for Body Sites at 6 Weeks
Description: as for outcome 41
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.075 (0.0160) | 0.100 (0.0171)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.185, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 41, analysis 1]; Least Squares Mean Difference = 0.025, 95% CI 2-sided [-0.012 to 0.062], Standard Error of Mean 0.0186

43. Secondary Outcome: Mean Stain Intensity for Body Sites at 8 Weeks
Description: as for outcome 41
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.063 (0.0166) | 0.112 (0.0184)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.014, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 41, analysis 1]; Least Squares Mean Difference = 0.049, 95% CI 2-sided [0.010 to 0.088], Standard Error of Mean 0.0196

44. Secondary Outcome: Mean Stain Area for Body Sites at 4 Weeks
Description: The facial and lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). The body regions were scored for area according to the following criteria. Stain area for the body of the tooth was scored as 0=no stain present, natural tooth color, 1=stain limited to pits and grooves; 2=stain outside pits/grooves, up to 10% of surface affected; 3=stain outside pits/grooves, over 10% of surface affected.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.064 (0.0133) | 0.056 (0.0145)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.623, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area for the body region and smoking status as covariates; Least Squares Mean Difference = -0.008, 95% CI 2-sided [-0.040 to 0.024], Standard Error of Mean 0.0160

45. Secondary Outcome: Mean Stain Area for Body Sites at 6 Weeks
Description: as for outcome 44
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.076 (0.0158) | 0.100 (0.0169)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.192, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area for the body region and smoking status as covariates; Least Squares Mean Difference = 0.024, 95% CI 2-sided [-0.013 to 0.061], Standard Error of Mean 0.0186

46. Secondary Outcome: Mean Stain Area for Body Sites at 8 Weeks
Description: as for outcome 44
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.067 (0.0180) | 0.124 (0.0200)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.009, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area for the body region and smoking status as covariates; Least Squares Mean Difference = 0.057, 95% CI 2-sided [0.014 to 0.099], Standard Error of Mean 0.0213

47. Secondary Outcome: Mean Stain Score for Facial Sites at 4 Weeks
Description: The mean stain score (0-9) per participant was determined by multiplying the individual area and intensity scores from each region and summing them then dividing by the number of sites scored. The facial surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). All four regions were scored for area and intensity according to the following criteria. Stain area for mesial, gingival, and distal regions were scored on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain covers entire area) and for the body of tooth on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain outside pits/grooves, over 10% of surface affected). The intensity of yellow-brown stains occurring in each region was assessed on a 4-point ordinal scale (0=no stain; 3=heavy, dark stain).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.063 (0.0314) | 0.058 (0.0342)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.893, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain score for the facial region and smoking status as covariates; Least Squares Mean Difference = -0.005, 95% CI 2-sided [-0.081 to 0.071], Standard Error of Mean 0.0384

48. Secondary Outcome: Mean Stain Score for Facial Sites at 6 Weeks
Description: as for outcome 47
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.118 (0.0399) | 0.140 (0.0427)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.655, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 47, analysis 1]; Least Squares Mean Difference = 0.021, 95% CI 2-sided [-0.073 to 0.116], Standard Error of Mean 0.0476

49. Secondary Outcome: Mean Stain Score for Facial Sites at 8 Weeks
Description: as for outcome 47
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.097 (0.0576) | 0.319 (0.0642)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 47, analysis 1]; Least Squares Mean Difference = 0.222, 95% CI 2-sided [0.084 to 0.359], Standard Error of Mean 0.0693

50. Secondary Outcome: Mean Stain Intensity for Facial Sites at 4 Weeks
Description: The facial surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). All four regions were scored for intensity according to the following criteria. The intensity of yellow-brown stains occurring in each region is unrelated to the area covered with stained pellicle. All four regions were assessed on a 4-point ordinal scale as 0=no stain, 1=faint stain (can be seen with close examination), 2=moderate stain (clearly visible and aesthetically unacceptable), 3=heavy, dark stain (obvious and aesthetically unacceptable).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.027 (0.0153) | 0.025 (0.0167)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.914, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain intensity for the facial region and smoking status as covariates; Least Squares Mean Difference = -0.002, 95% CI 2-sided [-0.039 to 0.035], Standard Error of Mean 0.0187

51. Secondary Outcome: Mean Stain Intensity for Facial Sites at 6 Weeks
Description: as for outcome 50
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.054 (0.0192) | 0.065 (0.0206)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.646, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 50, analysis 1]; Least Squares Mean Difference = 0.011, 95% CI 2-sided [-0.035 to 0.056], Standard Error of Mean 0.0229

52. Secondary Outcome: Mean Stain Intensity for Facial Sites at 8 Weeks
Description: as for outcome 50
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.042 (0.0257) | 0.144 (0.0286)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 50, analysis 1]; Least Squares Mean Difference = 0.102, 95% CI 2-sided [0.040 to 0.163], Standard Error of Mean 0.0309

53. Secondary Outcome: Mean Stain Area for Facial Sites at 4 Weeks
Description: The facial surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). All four regions were scored for area according to the following criteria. Stain area for mesial, gingival, and distal regions were scored as 0=no stain present, natural tooth color; 1=thin line of stain, may be discontinuous; 2=thick line or band of stain; 3=stain covers entire area and for the body of tooth as 0=no stain present, natural tooth color, 1=stain limited to pits and grooves; 2=stain outside pits/grooves, up to 10% of surface affected; 3=stain outside pits/grooves, over 10% of surface affected.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.032 (0.0147) | 0.033 (0.0160)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.930, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area for the facial region and smoking status as covariates; Least Squares Mean Difference = 0.002, 95% CI 2-sided [-0.034 to 0.037], Standard Error of Mean 0.0179

54. Secondary Outcome: Mean Stain Area for Facial Sites at 6 Weeks
Description: as for outcome 53
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.059 (0.0188) | 0.075 (0.0201)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.486, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 53, analysis 1]; Least Squares Mean Difference = 0.016, 95% CI 2-sided [-0.029 to 0.060], Standard Error of Mean 0.0224

55. Secondary Outcome: Mean Stain Area for Facial Sites at 8 Weeks
Description: as for outcome 53
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.047 (0.0281) | 0.160 (0.0313)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 53, analysis 1]; Least Squares Mean Difference = 0.112, 95% CI 2-sided [0.045 to 0.180], Standard Error of Mean 0.0338

56. Secondary Outcome: Mean Stain Score for Lingual Sites at 4 Weeks
Description: The mean stain score (0-9) per participant was determined by multiplying the individual area and intensity scores from each region and summing them then dividing by the number of sites scored. The lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). All four regions were scored for area and intensity according to the following criteria. Stain area for mesial, gingival, and distal regions were scored on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain covers entire area) and for the body of tooth on a 4-point ordinal scale (0=no stain present, natural tooth color; 3=stain outside pits/grooves, over 10% of surface affected). The intensity of yellow-brown stains occurring in each region was assessed on a 4-point ordinal scale (0=no stain; 3=heavy, dark stain).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.596 (0.0831) | 0.716 (0.0910)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.237, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain score for the lingual region and smoking status as covariates; Least Squares Mean Difference = 0.120, 95% CI 2-sided [-0.080 to 0.320], Standard Error of Mean 0.1006

57. Secondary Outcome: Mean Stain Score for Lingual Sites at 6 Weeks
Description: as for outcome 56
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.586 (0.0949) | 1.106 (0.1020)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 56, analysis 1]; Least Squares Mean Difference = 0.521, 95% CI 2-sided [0.298 to 0.743], Standard Error of Mean 0.1120

58. Secondary Outcome: Mean Stain Score for Lingual Sites at 8 Weeks
Description: as for outcome 56
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.677 (0.1146) | 1.244 (0.1283)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 56, analysis 1]; Least Squares Mean Difference = 0.567, 95% CI 2-sided [0.295 to 0.839], Standard Error of Mean 0.1367

59. Secondary Outcome: Mean Stain Intensity for Lingual Sites at 4 Weeks
Description: The lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). All four regions were scored for intensity according to the following criteria. The intensity of yellow-brown stains occurring in each region is unrelated to the area covered with stained pellicle. All four regions were assessed on a 4-point ordinal scale as 0=no stain, 1=faint stain (can be seen with close examination), 2=moderate stain (clearly visible and aesthetically unacceptable), 3=heavy, dark stain (obvious and aesthetically unacceptable).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.282 (0.0406) | 0.344 (0.0444)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.210, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain intensity for the lingual region and smoking status as covariates; Least Squares Mean Difference = 0.062, 95% CI 2-sided [-0.036 to 0.160], Standard Error of Mean 0.0491

60. Secondary Outcome: Mean Stain Intensity for Lingual Sites at 6 Weeks
Description: as for outcome 59
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.279 (0.0467) | 0.541 (0.0501)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 59, analysis 1]; Least Squares Mean Difference = 0.262, 95% CI 2-sided [0.153 to 0.372], Standard Error of Mean 0.0550

61. Secondary Outcome: Mean Stain Intensity for Lingual Sites at 8 Weeks
Description: as for outcome 59
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.314 (0.0549) | 0.596 (0.0614)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 59, analysis 1]; Least Squares Mean Difference = 0.281, 95% CI 2-sided [0.151 to 0.411], Standard Error of Mean 0.0654

62. Secondary Outcome: Mean Stain Area for Lingual Sites at 4 Weeks
Description: The lingual surfaces of the maxillary and mandibular anterior teeth (teeth #6-11 and #22-27) were scored using the Macpherson Modification of the Lobene Stain Index. Each surface was divided into 4 regions (gingival, mesial, distal, and body). All four regions were scored for area according to the following criteria. Stain area for mesial, gingival, and distal regions were scored as 0=no stain present, natural tooth color; 1=thin line of stain, may be discontinuous; 2=thick line or band of stain; 3=stain covers entire area and for the body of tooth as 0=no stain present, natural tooth color, 1=stain limited to pits and grooves; 2=stain outside pits/grooves, up to 10% of surface affected; 3=stain outside pits/grooves, over 10% of surface affected.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 47 | 45
units on a scale | 0.293 (0.0409) | 0.359 (0.0448)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.187, ANCOVA — The significance threshold level was 0.05 (two-sided); Terms included treatment as a factor and baseline mean stain area for the lingual region and smoking status as covariates; Least Squares Mean Difference = 0.066, 95% CI 2-sided [-0.033 to 0.165], Standard Error of Mean 0.0496

63. Secondary Outcome: Mean Stain Area for Lingual Sites at 6 Weeks
Description: as for outcome 62
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 44
units on a scale | 0.277 (0.0460) | 0.533 (0.0495)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 62, analysis 1]; Least Squares Mean Difference = 0.256, 95% CI 2-sided [0.148 to 0.364], Standard Error of Mean 0.0544

64. Secondary Outcome: Mean Stain Area for Lingual Sites at 8 Weeks
Description: as for outcome 62
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Number analyzed (Participants) | 46 | 41
units on a scale | 0.325 (0.0560) | 0.598 (0.0628)
Statistical Analysis 1: Comparison: Crest® Regular Toothpaste vs 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 62, analysis 1]; Least Squares Mean Difference = 0.273, 95% CI 2-sided [0.140 to 0.406], Standard Error of Mean 0.0669

ADVERSE EVENTS:
Time Frame: Week 8, +30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 4 (Week 8). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | Crest® Regular Toothpaste | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse)
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 3/48 | 2/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crest® Regular Toothpaste (N=48) | 11794-050 (1.5% Potassium Oxalate & pH 4.2 Mouth Rinse) (N=48)
Nasopharyngitis (Infections and infestations) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agreed not to publish the study results without prior sponsor approval.